CLINICAL TRIAL: NCT06088225
Title: Clinically Study the Ocular Axial Length and Sphere Equivalence Changes of Children With Distance-image Screen Usage for One Year
Brief Title: Myopia Preventing With Distance-image Screen
Acronym: DIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Airdoc Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Beijing Airdoc MPC Co., Ltd.
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Myopia, Progressive
Keywords: Myopia; children
MeSH Terms: conditions — Myopia, Degenerative; Myopia

STUDY DESIGN:
Intervention Model Description: Paired testing those ocular parameters before and after 12-month usage of distance-image screen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Distance -image screen (Experimental): Distance -image screen is a device to make image in the distance of 6-meters when reading and learning at near. The investigators will ask the subjects to use the distance - image screen for 12 month
  Interventions: Device: distance-image screen

INTERVENTIONS:
Device: distance-image screen — Distance-image screen is a screen make each image at distance of 6-meters to reduce the accommodation and convergence for eyes during the reading and learning with screens.

SUMMARY:
This study is for testing the efficacy and safety of distance-image screens for preventing myopia in children for 12 month. Each subjects would be asked to paired test the ocular parameters between before and after 12-month distance-image screens.

DETAILED DESCRIPTION:
This study is for testing the efficacy and safety of distance-image screens intended usage for preventing myopia in children with reading after a 6-meter-distant-image device. It was a prospective study. The investigators would like to recruit 100 volunteers, aged 6 years 16 in Beijing.

All the volunteers will be complete examined their ocular parameters before using the distant-image screen in a random order for at least 2 hours daily for 12 month. The changes of ocular axial length and refractive error were both calculated before and after 12-month usage for paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* (1) Must be 6~12 years old;
* (2) Must be best corrected visual acuity < logMAR: 0.1;
* (3) Spherical Equivalence (SE) must be -1.00~ + 6.00 Diopter (D),
* (4) Spherical Equivalence (SE) must have changed > 1.25 Diopter (D) in the recent 2 years;
* (5) Must be astigmatism <1.75 Diopter (D);
* (6) Must be anisometropia <1.75 Diopter(D).

Exclusion Criteria:

* (1) Strabismus disease;
* (2) Amblyopia disease;
* (3) Cataract disease;
* (4) Glaucoma disease;
* (5) Severe dry eye disease;
* (6) Cannot use distance-image screen for 12 month;
* (7) Other severe diseases that would effect the use of distance-image screen.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of ocular axial length (mm) | 12-month
  IntraOcularLens (IOL) master biometry will exam each eye before the testing and after the testing with distance-image screen
Changes of refractive error (D) | 12-month
  Cycloplegic refraction with autorefractor will test each eye before the testing and after the testing with distance-image screen

SECONDARY OUTCOMES:
Changes of center macular thickness (um) | 12-month
  Optic Coherent Topograph (OCT) of macular fovea central thickness will be made to compare the thickness before and after using distance-image screen
Changes of subretina choroidal thickness (um) | at 12-month
  Optic Coherent Topograph (OCT) with Enhanced Depth Imaging (EDI) scan of macular fovea central thickness will be done to compare the thickness before and after using distance-image screen
Changes of other regions choroidal thickness (um) | 12-month
  Optic Coherent Topograph (OCT) with Enhanced Depth Imaging (EDI) scan of other regions choroidal thickness will be done to compare the thickness before and after using distance-image screen

CONTACTS AND LOCATIONS:
Locations (1):
- Airdoc MPC Opthalmology Clinics, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No